CLINICAL TRIAL: NCT04323462
Title: Intensive Glycemic Control For Diabetic Foot Ulcer Healing: A Multicenter Randomized Control Study (IN-GLOBE Study)
Brief Title: Intensive Glycemic Control For Diabetic Foot Ulcer Healing
Acronym: INGLOBE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Collaborators: Institute of Post-Graduate Medical Education and Research, Kolkata (Other); Jawaharlal Institute of Postgraduate Medical Education & Research (Other Government); All India Institute of Medical Sciences, Bhubaneswar (Other)
Responsible Party: Principal Investigator, Ashu Rastogi, Assistant Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 100/20
Record Dates: First submitted 2020-03-23; First posted 2020-03-26 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Diabetic Foot Ulcer
Keywords: Diabetes; Intensive Glycemic Control; Diabetic Foot Ulcer; Wound Healing; HbA1c
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus | interventions — Insulin Glargine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigator and the Outcome assessor will not be aware of group allocation and the treatment thus offered.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive Glucose Control (Experimental): Intensive Glucose control Insulin ≥3 times per day; Goals: prePBG 80-130 & post PBG <180 (60% of all readings); HbA1c <8% at 3 months SMBG at least 14 readings/week (3-5 FBG, rest PPBG) and/or CGMS readings Reexamined weekly for 1 month; then fortnightly for 3 months and then monthly till 6 months
  Intensive subgroup will receive a standard glucometer with strips as one-week supply or CGMS for glycemic monitoring. They will receive a diabetic monitoring log/chart for home use. The chart and glucometer will have to be shown at each week of follow up. Number of hypoglycemic events in past week will be checked for each patient. This sub group will receive instructions to use 3 times bolus (regular/analogue) and single time basal insulin (glargine). Treatment goals will be conveyed at first contact and reinforced at each visit. Insulin dose modulation will be done telephonically. Patients will be reviewed weekly for 1 month and then fortnightly.
  Interventions: Drug: Insulin Glargine
- Conventional Glucose control (Active Comparator): Fixed dosage of oral anti-diabetic drugs/insulin per week as patient is receiving prior; Insulin <3 times per day SMBG <3 times per day
  Interventions: Drug: Diabetic DM

INTERVENTIONS:
Drug: Insulin Glargine — Three times bolus insulin with regular or Shorter acting insulin
  Other Names: Bolus Insulin
  Arms: Intensive Glucose Control
Drug: Diabetic DM — Previously receiving OADs and/or basal insulin
  Other Names: OADs
  Arms: Conventional Glucose control

SUMMARY:
With the available molecular and cellular evidence of impaired wound healing due to hyperglycemia, investigators postulate hypothesis asking whether intensive glycemic control could improve diabetic foot ulcer healing rates. A study showed improvement in phagocytic activity of macrophages after 5 days of intensive glycemic improvement in 21 patients of diabetes. Another retrospective cohort study studied the effect on HbA1c as predictor of healing rate in DFU. Latter found significant association of HbA1c with wound area healing rate. However a recent systematic review failed to find any randomized control trial comparing the effect of intensive versus conventional glycemic control for treating DFU. Hence, investigators want to explore the hypothesis by conducting a randomized control trial with the primary aim of wound healing in patients of diabetic foot ulcer in response to intensive glycemic control in comparison to conventional glycemic management.

DETAILED DESCRIPTION:
BURDEN OF DIABETIC FOOT According to International Diabetic Federation, there will be over 642 million people with diabetes in the world by 2040.Diabetic Foot Ulcer (DFU) is one of the most serious, most costly and at times life threatening complication of diabetes. The lifetime incidence of foot ulcer occurrence in diabetes is up to 25%. Both prevalence and incidence of DFU is higher in developing countries due to multitude of factors like poverty, poor sanitation & hygiene, barefoot walking, lack of education, poor healthcare access.

DFU related morbidity and hospitalization has shown a meteoric rise. One study showed that 20% of admissions in patients of diabetes were due to DFU. 56%of ulcers become infected and 1 in 5 of these will requiresome level of amputation.In addition, it has been projected that 15% of diabetic foot ulcers result in lowerextremity amputations and 85% of diabetic patientswho undergo lower extremity amputations had an ulcerprior to amputation.The 5-year relative mortality afterdiabetic foot ulcer is 48%, second only to lung cancer.

Multiple risk factors have been attributed to the development of DFU including male gender, duration of diabetes >10 years, older age, diminished vision, peripheral vascular disease, high BMI, sensory neuropathy, retinopathy, nephropathy, HbA1c, foot deformity, high plantar pressures, poor foot care habits, barefoot walking etc. From DCCT there exists robust evidence that strict glycemic control can decrease all diabetic related complications. There are other studies demonstrating improvements in neuropathy and peripheral vascular disease as a result of strict glycemic control. However, there is no specific evidence/intervention for DFU prevention.

IMPAIRED WOUND HEALING IN DIABETES Wound healing is impaired in diabetes at multiple stages. The defects are observed at both cellular and molecular levels. Extrinsic factors like mechanical stress, trauma and ischemia negatively influence the healing process. Hyperglycemia itself has been shown to have deleterious effect on wound healing through formation of advanced glycation end products (AGEs) & reactive oxygen species (ROS) which induce the production of inﬂammatory molecules (TNF-α, IL-1) and interfere with collagen synthesis. There is interference in collagen synthesis due to increased expression of matrix metalloproteinases.

CHALLENGES WITH RESEARCH IN THIS AREA With the clinical benchmarks set by major trials like UKPDS, it is often difficult for clinicians to ethically conduct any study investigating the effects of intensive versus conventional glycemic control. Even on demonstrating the clinical benefit involving intensive glycemic control, it is a difficult task to recruit as well as follow up subjects. Many diabetic patients are frail and have multiple co-morbidities that render them incapable of following such interventions. Intensive glycemic control makes these individuals prone to the detrimental effects of hypoglycemia. In a trial investigating the effect of hyperglycemia and intensive glycemic control on DFU healing, the authors faced many challenges in recruiting and allocating the patients. This trial was completed without any results.

There is marked variation in the definition of intensive glycemic control between guidelines and trials.Most of the current glycemic targets for diabetes are based onseveral pioneering trials that investigated the effects of intensiveglycemic control compared to conventional treatments. Importantly, the beneficial effects on microvascular complicationsfrom using intensive glycemic control took more than five yearsto emerge, and the benefits were less pronounced for people withadvanced type 2 diabetes compared to those with new-onset type2 diabetes. Nevertheless, diabetic foot ulcer specific outcomes were not studied or neglected in these trials. Hence, the onus is on new investigators to study the outcomes in DFU through the prism of intensive glycemic control.

In many trials investigating intensive versus conventional glycemic control,lower limb amputation was an outcome measure. This outcome was not reported in relation to presentation with, development of, or healing of foot ulceration. Amputation was due to the ease of measurement and definitive nature of such a practical end-point. However, there are inconsistencies in the true estimation of amputation as an outcome. The UKPDS defined amputation as a major limbcomplication requiring lower limb amputation of a digit or anylimb for any reason and included digital amputations which areusually classified as minor amputations. A Cochrane review concluded that intensive glucose control reduced the risk of amputation by 36% in type 2 diabetes (RR 0.64, 95% CI: 0.43 to 0.95; 6960 participants ineight trials). However, this information was based on amputations defined in several ways (including both minor and major amputations). Although this data provides evidence to endorse the efficacy of intensive glycemic control in preventing amputations, its exact correlation to foot ulcer healing remains unanswered.It is a known fact that foot ulceration often precedes amputation, therefore, ulcer specific measures like time to ulcer healing, percent reduction in ulcer area, need to be measured as an outcome. From a patient and HRQoL point of view, foot ulcer healing can be seen as a beneficial outcome over a damaging endpoint like amputation.

In a meta-analysis of the six control arms ofwound-healing trials in patients with a neuropathic ulcer, 24% of the ulcers were healed at 12 weeks and only 31%at 20 weeks. But these data were likely influenced by selection bias, as the elderly patient with multiple co-morbidities is usually excluded from such trials, follow-up was short and treatment was suboptimal and non- EVIDENCE OFNEED FOR INTENSIVE GLYCEMIC CONTROL IN DFU Various studies highlighting the importance of hyperglycemia and glycemic control in diabetic foot ulcer healing are described below.

In a multi-center study, poor glycemic (blood glucose) control was evident in nearly half of the participants who had foot ulcers, with 49% having an HbA1c (glycemic measure) level above 8.4%.

In a retrospective cohort study of 183 diabetic patients conducted at the John Hopkins Wound Center, it was seen that HbA1c was an important clinical predictor of the rate of wound healing. The mean HbA1c was 8.0%. For each 1%-point increase in HbA1c level,the daily wound healing ratedecreased by 0.028 cm² per day (95% CI: 0.003 to 0.054). This was irrespective of presence of neuropathy (n=109), smoking status (n=121) and peripheral arterial disease (n=53). The study didn't throw any light on anti-diabetic treatment received by patients.

In another retrospective study of 63 diabetic patients conducted at a Midwestern outpatient wound care clinic in USA for 3 years, it was seen that the HbA1c values closest to ulcer closure ranged from 5.3 to12.3 (mean, 7.68 [SD, 1.81]). It was also found that patients with higher HbA1c levels did experience wound healing, but in a significantlylonger period than those with lower HbA1c. Approximately 80% of this sample (n = 50)had peripheral vascular disease, and more than 60% (n = 39) hadrenal disease. Here also the investigators didn't mention the anti-diabetic treatment being received by patients.

An Indian prospective study (over 2 years) has explored the concept of HbA1c as a predictor of healing rate in diabetic ulcers. 100 diabetic patients were equally divided into 2 groups with mean HbA1c levels of 6.50 ± 0.441 in Group A and Group B with the mean value of 10.40 ± 1.550. Subsequently, standard treatment protocols were followed, and mean reduction in ulcer area, length, and width were measured; a statistically significant difference was found in the mean area change per day between the two groups with P<0.0001. However, the study did not explore the effect of intensive glycemic treatment in the uncontrolled diabetic subgroup.

Investigators in Barcelona, Spain addressed the issue of impairment in phagocytic activity in relation to glycemic control and, whether or not this impairment could be reversible after improving blood glucose levels. In their case control study, 21 type 2 DM and 21 healthy volunteers were prospectively recruited. Baseline HbA1c was 8.78 ± 2.01 in T2DM patients whereas it was 5.79 ± 0.45 in healthy volunteers. Baseline FBG was 9.49 ± 3.15 in T2DM patients whereas it was 5.73 ± 0.83 in healthy volunteers. By use of flow cytometry they were able to deduce that Type 2 diabetic patients showed a lower percentage of activated macrophages in comparison with non-diabetic subjects (54.00618.93 vs 68.53612.77%; p = 0.006). Also,significant negative correlations between phagocytic activity and fastingglucose (r = 20.619, p = 0.004) and HbA1c (r = 20.506, p = 0.019) were detected. In their intervention study 12 previous T2DM patients were admitted and treated intensively (9-point blood glucose profile) for 5 days. In these patients who underwent metabolic optimization, a significant increase in phagocytic activitywas observed (p = 0.029). The investigators postulated that the reversibility of phagocytosis dysfunction after a short period of glycemic control may have been attributable not only to the normalization of the diabetic milieu but also to the effect of exogenous insulin.

Another prospective study conducted in Oregon, USA investigated whether different diabetic treatment regimens affect diabetic foot ulcer healing. In this study 85 patients were followed up for a period of 2 years. Insulin treatment was apart of diabetes management in 52 (61.2%) cases. Insulin therapy significantly increased thewound healing rate (30.3% [20/66 ulcers] vs. 9.8% [4/41 ulcers]) (p=0.013). In multivariaterandom-effect logistic regression model, adjusting for age, gender, smoking status, type of diabetes, hypertension, chronic kidney disease, peripheral arterial disease, oral hypoglycemic use, wound infection, involved side, presence of Charcot's deformity, gangrene, osteomyelitis on x-ray, and serum hemoglobin A1C levels, insulin treatment was associated with a higher chance of complete healing (beta±SE: 15.2±6.1, P=0.013).

In a Cochrane systematic review aimed to assess the effects of intensive glycemic control compared to conventional control on the treatment of foot ulcers in people with type 1 and type 2 diabetes. The authors searched for evidence in both published and unpublished material. They were unable to find any clinical trials which had successfully investigated the impact of intensive versus conventional glycemic control on foot ulcer outcomes. Investigators want to fill this lacuna by conducting a randomized control trial with the primary aim of wound healing in participants of diabetic foot ulcer on intensive glycemic control versus conventional treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years
2. Patients of DM according to ADA guidelines
3. HbA1c >8% (single occasion at screening) and/or FBG >130 on 3 consecutive occasions
4. DFU: Wagner grade 1, 2 & 3 or UTS 1, 2-3B
5. Duration of ulcer>2 weeks
6. Wound size: >1cm2
7. Willingness to sign consent form & participate in the study
8. Capacity to attend visits at hospital for review

Exclusion Criteria:

1. Diagnosis with unpredictable healing ability e.g. malignancy, depression, HIV, CTD, steroid use
2. Dialysis requiring CKD & eGFR <30 ml/min
3. Anemia with hemoglobin <10 gm/dl
4. Active Charcot foot
5. PEDIS 4: life threatening DFU
6. Pregnancy
7. ABI <0.7
8. Refusal to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Wound Healing | 12 weeks
  Number of wounds that have closed Completely in the two arms. Complete closure of wound will be defined as epithelial action of ulcer

SECONDARY OUTCOMES:
wound area | 4 and 12 weeks
  reduction in Wound Area in cm2 from baseline . The ulcer area will be measured in two dimensions with an automated camera with the provision of correction and drawing of ulcer margins by the investigator.
time to ulcer healing | upto 12 weeks
  Time to healing of ulcer in weeks from baseline

OTHER OUTCOMES:
amputation | 12 weeks
  Number of amputations

CONTACTS AND LOCATIONS:
Locations (2):
- India (2):
  - IPGMER, Kolkata, West Bengal
  - Deptt of Endocrinology, Chandigarh

IPD SHARING:
Plan to Share IPD: No
The Individual data of participants will not be shared amongst investigators. However, it will be anonymously entered into electronic database.